CLINICAL TRIAL: NCT00261378
Title: Prospective Randomised Study of Doxorubicin in the Treatment of Hepatocellular Carcinoma by Drug-Eluting Bead Embolisation (PRECISION V)
Brief Title: Prospective Randomised Study of Doxorubicin in the Treatment of Hepatocellular Carcinoma by Drug-Eluting Bead Embolisation
Acronym: PRECISIONV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA1008
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Primary Liver Cancer
Keywords: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Transarterialchemoembolisation (TACE) (Active Comparator): Conventional TACE with doxorubicin
  Interventions: Device: Transarterialchemoembolisation (TACE)
- DC Bead (Other): DC Bead with doxorubicin
  Interventions: Device: DC Bead with Doxorubicin

INTERVENTIONS:
Device: Transarterialchemoembolisation (TACE)
  Other Names: Conventional TACE with doxorubicin
  Arms: Transarterialchemoembolisation (TACE)
Device: DC Bead with Doxorubicin
  Arms: DC Bead

SUMMARY:
The objective of this study is to assess the safety and efficacy of DC Bead™ delivered by intra-arterial embolisation for the treatment of Hepatocellular Carcinoma

ELIGIBILITY:
Inclusion criteria

* Patients with a confirmed diagnosis of HCC according to the EASL criteria for diagnosis, see appendix 4 and staged according to the BCLC criteria.
* Patient chooses to participate and has signed the informed consent document
* Age above 18 years old
* Patients with HCC not suitable for resection or percutaneous ablation according to the BCLC Staging classification, see Figure 2.
* Patient is eligible for resection or percutaneous ablation but the treatment is unfeasible or the patient has declined. This decision must be documented in the patient's records.
* Patient is eligible for chemoembolisation prior to transplantation and the expected transplant waiting time exceeds 6 months.
* Patients who demonstrates recurrence following potentially curative treatment (resection and percutaneous ablation) who have clearly measurable disease according to RECIST or EASL
* Patients with Performance Status ECOG 0 and 1
* Patients with well preserved liver function (Child-Pugh A and B)
* Patients with bilobar disease who can be treated superselectively in a single session or both lobes able to be treated within 3 weeks.

Exclusion criteria

* Patients with another primary tumour, with the exception of conventional basal cell carcinoma or superficial bladder neoplasia
* Patients previously treated with transarterial embolisation (with or without chemotherapy).
* Patients previously treated with anthracyclines (ie doxorubicin).
* Patients' whose only measurable disease is within an area of the liver previously subjected to radiotherapy.
* Advanced liver disease:

  * Child-Pugh C,
  * active gastrointestinal bleeding,
  * encephalopathy or clinically relevant ascites.
* Bilirubin levels >3mg/dl
* Advanced tumoural disease:

  * BCLC class C, (vascular invasion including segmental portal obstruction, extrahepatic spread or cancer-related symptoms= ECOG 2, 3 and 4) or
  * BCLC class D (WHO performance status 3 or 4, Okuda III stage) or
  * Diffuse HCC defined as >50% tumour involvement of the whole liver
* Any contraindication for doxorubicin administration:

  * serum bilirubin >5mg/dL,
  * WBC <3000 cells/mm3
  * neutrophil <1500 cells/mm3,
  * cardiac ejection fraction <50 percent assessed by isotopic ventriculography, echocardiography or MRI
* Any contraindication for hepatic embolisation procedures:

  * porto-systemic shunt,
  * hepatofugal blood flow;
  * impaired clotting tests (platelet count <50000/mm3, prothrombin activity <50 percent),
  * renal insufficiency/failure, serum creatinine > 2mg/dl (177umol/l)
  * severe atheromatosis,
  * AST and/or ALT >5x ULN or, when greater >250U/l
* Women who are pregnant or breast feeding
* Allergy to contrast media
* Contraindication to hepatic artery catheterisation, such as severe peripheral vascular disease precluding catheterisation
* The availability of alternative therapies those, in the judgment of the physician (referring or treating), are more appropriate for the patient
* Any co-morbid disease or condition or event that, in the investigator's judgment, would place the patient at undue risk, that would preclude the safe use of DC Bead™, or TACE
* Patients who are contraindicated for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2005-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate measured according to RECIST and EASL | 6 months

SECONDARY OUTCOMES:
Toxicity | 6 month
Change in Alpha Fetal Protein (AFP) over time | 6 months
Time to hospital discharge | 6 months
Safety | 6 months
Other procedures or interventions required | 6 months
Cardiotoxicity | 6 months
Local Tumour Response | 6 months
Health care resource use | 6 months
Patient quality of life | 6 months
Time To Progression | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof Johannes Lammer, Principal Investigator — The Allgemines Krankenhaus, Vienna, 1090, Austria
Locations (17):
- Austria (2):
  - Medizinische Universitat Innsbruck, Innsbruck
  - Allgemines Krankenhaus Vienna, Vienna
- France (7):
  - L'Hopital Beaujon, Clichy
  - Hopital Claude Huriez, Lille
  - Groupement Hospitalier Edouard Herriot, Lyon
  - Hopital Archet II, Nice
  - Hopital Pitie Salpetriere, Paris
  - CHU Rangueil, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Klinikum der Johann-Wolfgang-Goethe-Universitat, Frankfurt am Main
  - Medicinische Hochschule Hannover, Hanover
  - Klinikum der Johannes Guttenberg, Mainz
  - Fakultat fur Klinische Medizin Mannheim Universitat, Mannheim
- Switzerland (4):
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Universitatsspital Zurich, Zurich

REFERENCES:
- [Derived] Vogl TJ, Lammer J, Lencioni R, Malagari K, Watkinson A, Pilleul F, Denys A, Lee C. Liver, gastrointestinal, and cardiac toxicity in intermediate hepatocellular carcinoma treated with PRECISION TACE with drug-eluting beads: results from the PRECISION V randomized trial. AJR Am J Roentgenol. 2011 Oct;197(4):W562-70. doi: 10.2214/AJR.10.4379. PMID 21940527